CLINICAL TRIAL: NCT05374161
Title: Efficacy of a Brief Intervention for Female Breast CANcer Based on Acceptance and Commitment Therapy (I-CAN-ACT) for Depression and Physical Pain: A 2-Arm Randomized Clinical Trial
Brief Title: An Intervention for Female Breast CANcer: Acceptance and Commitment Therapy (I-CAN-ACT) for Depression and Physical Pain
Acronym: I-CAN-ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Maria Karekla, Associate Professor, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K3_K1_2
Record Dates: First submitted 2022-01-04; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Female Breast Cancer; Depression; Pain
Keywords: Female Breast Cancer; Physical Pain; Depression; Quality of Life; Brief ACT-based Intervention; RCT
MeSH Terms: conditions — Depression; Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: A 2-arm RCT will be conducted (brief ACT-based intervention vs waitlist control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief ACT-based intervention (Experimental): A 6- week ACT intervention for depression and physical pain will be delivered.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Waitlist control group (WL) (Other): The WL control group will receive treatment as usual, just like women in the experimental condition.
  Interventions: Other: Waitlist Control Group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The ACT-based intervention will be delivered in a group format. Due to the COVID-19 pandemic and given that breast cancer patients are considered a vulnerable population, the intervention will be administered online through a GDPR compliant platform. The six, weekly, 90-minute treatment sessions (total of 9 hours) will be conducted in groups of approximately 8-10 participants and one therapist.
  Arms: Brief ACT-based intervention
Other: Waitlist Control Group — Participants randomized to the WL condition will be asked to continue receiving the services they receive from anti-cancer associations (receiving care from nurses, or/and support from social workers, or/and physiotherapy or/and individual psychological support from licensed psychologists just like the women in the experimental condition).
  Arms: Waitlist control group (WL)

SUMMARY:
As a result of the cancer diagnosis and medical therapies, women with breast cancer often encounter debilitating cooccurring psychological and physical symptoms. While pain constitutes one of the most common adverse physical side effects of medical treatment reported by breast cancer patients, the most prevalent psychological symptom they seek psychological help for is depressive symptoms. Acceptance and Commitment Therapy (ACT) in psychosocial oncology care may be particularly beneficial in targeting depression and cancer-related pain. The aim of the I-CAN-ACT project is to examine in a RCT the efficacy of a brief ACT-based intervention for both depression and physical pain (6 online sessions) compared to a waitlist control on various outcomes in women with breast cancer. Outcomes will include quality of life, physical pain intensity and interference, depression, and anxiety in women with breast cancer. These will be assessed at post-treatment and at the 1-month, 3-month, 6-month and 1 year follow-ups (for Marianna Zacharia's PhD thesis, results will be presented until the 3-month follow-up). Also, the Acceptability and Feasibility of the intervention will be assessed. That is, participants' treatment acceptability and adherence to the brief ACT intervention in terms of retention, treatment engagement and satisfaction with each session and with the overall treatment will be assessed. Participants' reasons for dropout will be recorded.

DETAILED DESCRIPTION:
As a result of the cancer diagnosis and medical therapies, women with breast cancer often encounter debilitating cooccurring psychological and physical symptoms. While pain constitutes one of the most common adverse physical side effects of medical treatment reported by breast cancer patients, the most prevalent psychological symptom they seek psychological help for is depressive symptoms. Acceptance and Commitment Therapy (ACT) in psychosocial oncology care may be particularly beneficial in targeting depression and cancer-related pain. The aim of the I-CAN-ACT project is to examine in a RCT the efficacy of a brief ACT-based intervention for both depression and physical pain (6 online sessions) compared to a waitlist control on various outcomes in women with breast cancer.

Based on preliminary empirical findings, the hypotheses of this study are:

1. The group ACT-based intervention will demonstrate significantly greater improvements in the primary outcome (quality of life: physical well-being, emotional well-being, social/family well-being, functional well-being, additional concerns for breast cancer) compared to the WL at post-treatment, at 1-month and 3-month follow-ups.
2. The group ACT-based intervention will demonstrate significantly greater reductions in the secondary outcomes (pain intensity and interference, depression and anxiety) compared to the WL at post-treatment, at 1-month and 3-month follow-ups.
3. The group ACT-based intervention will present significant improvements in the ACT components (acceptance, cognitive defusion, contact with the present moment, self-as-context, self-compassion, values clarification, committed action) compared to the WL at post-treatment, at 1-month and 3-month follow-ups.
4. It is hypothesized that the mechanisms/core processes, via which ACT is expected to exert its effects, will mediate pre to 1-month follow-up and pre to 3-month follow-up quality of life scores (primary outcome) for the ACT-based intervention.
5. It is hypothesized that the mechanisms/core processes, via which ACT is expected to exert its effects, will mediate pre to 1-month follow-up and pre to 3-month follow-up scores of secondary outcomes (physical pain intensity and interference, depression, anxiety).
6. Completing any ACT skill in a session will lead to improvement in that specific skill (ACT proposed mechanism of action) in-the-moment within each week of the group ACT-based intervention.

This is the first study to:

i. examine the longitudinal effects (1-month and 3-month follow ups) of an ACT intervention on both depression and physical pain, which often co-occur in female breast cancer patients ii. examine all the processes of change in ACT responsible for effective treatment outcomes in women with breast cancer iii. offer a brief ACT intervention for this population iv. assess participants' treatment acceptability and adherence to an ACT-based intervention in terms of retention, treatment engagement and satisfaction with treatment for this population v. assess therapists' fidelity/adherence to the protocol and the ACT approach as well as the therapists' competence, when implementing a RCT for women with breast cancer vi. employ the innovative methodological approach of Ecological Momentary Assessment through a mobile application in addition to standardized pre post-follow-up self-report questionnaires to assess changes in the ACT processes as a result of intervention

ELIGIBILITY:
Inclusion Criteria:

* Understanding and speaking fluently in Greek
* Age 18 and older
* Education level should be at least elementary school (ability to read and write)
* Diagnosed breast cancer in stages I, II or III
* Underwent breast surgery
* Experiencing at least mild depression and at least mild intensity and interference of physical pain

Exclusion Criteria:

* A history of metastasis (stage IV cancer)
* Significant cognitive impairment assessed using the Mini-mental State Examination (MMSE score < 20)
* A history of severe psychopathology (i.e., psychosis), suicidal ideation, substance use problems before breast cancer

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with breast cancer
Enrollment: 88 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Functional Assessment of Cancer Therapy - Breast (FACT-B; Brady et al., 1997) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  It consists of five well-being domains: physical well-being (7 items), emotional well-being (6 items), social/family well-being (7 items) and functional well-being (7 items), which constitute the Functional Assessment of Cancer Therapy - General (FACT-G; Cella et al., 1993) and the additional concerns for breast cancer, the Breast Cancer Subscale (BCS; 10 items). Each item on the FACT-B is rated on a five-point scale ranging from 0 = "not at all" to 4 = "very much". The total score can range from 0 to 144 and is the sum of scores from all five subscales. Higher scores reveal greater perceived quality of life.

SECONDARY OUTCOMES:
Change in the Hospital Anxiety and Depression Scale (HADS; Greek version: Mystakidou et al., 2004 and Michopoulos et al., 2008; English version: Zigmond & Snaith, 1983) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  It is a 14-item self-report measure of psychological distress in individuals with physical health problems (Johnston, Pollard, & Hennessey, 2000; Roberts, Bonnici, Mackinnon, & Worcester, 2001). Scale scores are thought to be unbiased by the existence of bodily illness (Zigmond & Snaith, 1983). HADS assesses anxiety (7 items) and depression (7 items) independently, rated on a four-point scale (range= 0-3; different anchors per item), with scores ranging between 0 and 21 per subscale. Higher scores indicate higher levels of anxiety and depression.
Change in the Brief Pain Inventory (BPI; Cleeland, 1989) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  It was initially developed in English in the USA (Cleeland, 1989) and has been validated in several languages. The Greek Brief Pain Inventory- Short Form (G-BPI; Mystakidou et al., 2001) is a 9-item self-report questionnaire used to assess pain intensity and pain interference in cancer patients. Patients are requested to rate their worst, least, average and current pain intensity and report current medications/treatment along with their perceived effectiveness on a 10-point scale, ranging from 0 = "no pain" to 10 = "pain as bad as you can imagine". Also, they are asked to rate the extent to which pain interferes with general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life on a 10-point scale, ranging from 0 = "does not interfere" to 10 = "completely interferes". Higher scores indicate higher pain intensity and higher pain interference.
Change in the Psyflex (Gloster et al., 2021) | A mobile application will be used, which will prompt the patients in the ACT intervention to answer the eight items of the PsyFlex. These prompts will take place twice per day for the six weeks of the intervention (Ecological Momentary Assessment).
  The PsyFlex (Gloster et al., 2021) is an 8-item self-report measure that assesses all six processes/skills of the ACT Hexaflex; that is psychological flexibility. Items of the PsyFlex are rated on a 5-point Likert type scale, ranging from 1 "very often" to 5 "very rarely". Higher scores indicate lower levels of psychological flexibility.
Change in the Greek Acceptance and Action Questionnaire - II (AAQ-II; Greek version: Karekla & Michaelides, 2017; English version: Bond et al., 2011) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The Greek Acceptance and Action Questionnaire - II (AAQ-II; Greek version: Karekla & Michaelides, 2017; English version: Bond et al., 2011) is a 7-item self-report measure of experiential avoidance or its reverse, psychological flexibility. Items are rated on a 7-point Likert scale, ranging from 1 = "never true" to 7 = "always true". Higher scores indicate greater experiential avoidance while lower scores indicate greater psychological flexibility.
Change in the Cognitive Fusion Questionnaire (CFQ; Greek version: Zacharia et al., 2021; English version; Gillanders et al., 2014) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The Cognitive Fusion Questionnaire (CFQ; Greek version: Zacharia et al., 2021; English version: Gillanders et al., 2014) is a brief, 7-item self-report scale of cognitive fusion. Items are rated on a 7-point Likert scale (range from 1 = "Never true" to 7 = "Always true". Higher scores indicate higher levels of cognitive fusion.
Change in the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R; Feldman, Hayes, Kumar, Greeson, & Laurenceau, 2007) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The Cognitive and Affective Mindfulness Scale-Revised (CAMS-R; Feldman, Hayes, Kumar, Greeson, & Laurenceau, 2007) is a 12-item self-report measure of mindfulness, designed based on the definition of mindfulness as "the awareness that emerges through paying attention on purpose, in the present moment, and non-judgmentally to the unfolding of experience moment to moment" (Kabat-Zinn, 2003, p. 145). Items are rated on a 4-point Likert scale, ranging from 1 "rarely/not at all" to 4 "almost always". Authors suggest the use of a total score.
Change in the Self-as-Context Scale (SACS; Zettle et al., 2018) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The Self-as-Context Scale (SACS; Zettle et al., 2018) is a brief (10-item) self-report scale of contextual self. Items are rated on a 7-point Likert scale, ranging from 1 "Strongly disagree" to 7 "Strongly Agree". Higher scores indicate higher levels of Centering, Transcending and Contextual Self.
Change in the Valuing Questionnaire (VQ; Smout, Davies, Burns, & Christie, 2014) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The Valuing Questionnaire (VQ; Smout, Davies, Burns, & Christie, 2014) is a 10-item measure that assesses the degree to which the person lives and acts in accordance to his/her values. Items are rated on a 7-point Likert type scale, ranging from 0 "never true" to 6 "always true".
Change in the Committed Action Questionnaire (CAQ; McCracken et al., 2015) | pre-treatment, mid-intervention assessment, post-treatment, 1-month follow-up, 3-month follow-up
  Committed Action Questionnaire (CAQ; McCracken et al., 2015), is an 8-item scale that examines goal-directed behaviors. Items are rated on a 7-point Likert-type scale, ranging from 0 "never true" to 6 "always true". Negatively worded items are reverse scored in order to indicate higher levels of committed actions. Higher scores indicate a higher tendency to persist in value-driven actions.
Change in the Self-Compassion Scale (SCS; English version: Neff, 2003; Greek version: Mantzios, Wilson, & Giannou, 2015) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The Self-Compassion Scale (SCS; English version: Neff, 2003; Greek version: Mantzios, Wilson, & Giannou, 2015) is a 26-item scale that measures six constituents of self-compassion. Items are rated on a 5-point Likert-type scale, ranging from "Almost Never" to "Almost Always". A total self-compassion score is calculated after reversing the negative subscale items and adding all subscale scores. Higher scores indicate higher self-compassion.
Change in The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Fatigue (EORTC QLQ-FA12; Weis et al., 2017) | pre-intervention, mid-intervention assessment (at the end of week 3), post-intervention (at 6 weeks), 1-month follow-up, 3-month follow-up
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Fatigue (EORTC QLQ-FA12, abbreviated as FA12) will be used as a measure of cancer related fatigue (Weis et al., 2017). It is comprised of 12 items, with four response categories for each item, coded with values from 1 to 4. Higher scores indicate greater fatigue.

OTHER OUTCOMES:
ACT Fidelity Measure (ACT-FM; O'Neill, Latchford, McCracken, & Graham, 2019) | The research assistant will be asked to complete the ACT-FM at the end of each of the six sessions.
  Therapists' ACT-consistent and ACT-inconsistent responses and behaviors will be assessed using the ACT Fidelity Measure (ACT-FM; O'Neill, Latchford, McCracken, & Graham, 2019). ACT-FM is a 25-item scale, which captures four important areas within ACT: Therapist Stance, Open Response Style, Aware Response Style and Engaged Response Style. The items are scored to measure the therapist's behaviors as consistent and inconsistent with these four areas. Items are rated on a range of 0 when the behavior did not occur to 3 when the behavior occurred extensively. Higher scores are assigned when the behavior occurs more consistently. A Total ACT Consistency Score (0-36) and a Total ACT Inconsistency Score (0-36) will be calculated for each session.
Change in the Session Rating Scale Version 3 (SRS V.3; Duncan et al., 2003) | Participants will be asked to complete the SRS V.3 after the end of each of the six sessions.
  The Session Rating Scale Version 3 is used on a session by session basis to assess the working alliance (SRS V.3; Duncan et al., 2003). The SRS V.3 entails four 10-cm visual analog scales, where participants are required to make a hash mark on a continuum line, which on the left represents the least satisfaction, and on the right represents the most satisfaction.
Treatment Acceptability and Adherence: Treatment Acceptability/Adherence Scale (TAAS; Milosevic, Levy, Alcolado, & Radomsky, 2015) | post-intervention (at 6 weeks)
  Overall participants' acceptability and adherence to treatment will be assessed with the Treatment Acceptability/Adherence Scale (TAAS; Milosevic, Levy, Alcolado, & Radomsky, 2015), a 10-item self-report scale. The scale is rated on a 7-point Likert scale, ranging from 1 "Disagree strongly" to 7 "Agree strongly". Six items are reversed when scoring (3, 4, 5, 7, 8 and 10) and scores may range from 10 to 70. Higher scores represent greater acceptability of treatment and greater ability to adhere to it.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Karekla, Ph.D., Principal Investigator — ACThealthy Lab, University of Cyprus
Locations (1):
- University of Cyprus, Nicosia, Non-US/Non-Canadian, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Cleeland, C. S. (1989). Measurement of pain by subjective report. Advances in Pain Research and Therapy, 12, 391-403.
- [Background] Duncan, B. L., Miller, S. D., Sparks, J. A., Claud, D. A., Reynolds, L. R., Brown, J., & Johnson, L. D. (2003). The Session Rating Scale: Preliminary psychometric properties of a "working" alliance measure. Journal of Brief Therapy, 3(1), 3-12.
- [Background] Feldman, G., Hayes, A., Kumar, S., Greeson, J., & Laurenceau, J. P. (2007). Mindfulness and emotion regulation: The development and initial validation of the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Journal of Psychopathology and Behavioral Assessment, 29(3), 177-190. https://doi.org/10.1007/s10862-006-9035-8
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Gloster, A. T., Block, V. J., Klotsche, J., Villanueva, J., Rinner, M. T., Benoy, C., ... & Bader, K. (2021). Psy-flex: A contextually sensitive measure of psychological flexibility. Journal of Contextual Behavioral Science, 22, 13-23. https://doi.org/10.1016/j.jcbs.2021.09.001
- [Background] Kabat-Zinn, J. (2003). Mindfulness-based stress reduction (MBSR). Constructivism in the Human Sciences, 8(2), 73-83.
- [Background] Karekla, M., & Michaelides, M. P. (2017). Validation and invariance testing of the Greek adaptation of the Acceptance and Action Questionnaire-II across clinical vs. nonclinical samples and sexes. Journal of Contextual Behavioral Science, 6(1), 119- 124. https://doi.org/10.1016/j.jcbs.2016.11.006
- [Background] Mantzios, M., Wilson, J. C., & Giannou, K. (2015). Psychometric properties of the Greek versions of the self-compassion and mindful attention and awareness scales. Mindfulness, 6(1), 123-132. https://doi.org/10.1007/s12671-013-0237-3
- [Background] McCracken LM, Chilcot J, Norton S. Further development in the assessment of psychological flexibility: a shortened Committed Action Questionnaire (CAQ-8). Eur J Pain. 2015 May;19(5):677-85. doi: 10.1002/ejp.589. Epub 2014 Sep 2. PMID 25181605
- [Background] Michopoulos I, Douzenis A, Kalkavoura C, Christodoulou C, Michalopoulou P, Kalemi G, Fineti K, Patapis P, Protopapas K, Lykouras L. Hospital Anxiety and Depression Scale (HADS): validation in a Greek general hospital sample. Ann Gen Psychiatry. 2008 Mar 6;7:4. doi: 10.1186/1744-859X-7-4. PMID 18325093
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Mystakidou K, Mendoza T, Tsilika E, Befon S, Parpa E, Bellos G, Vlahos L, Cleeland C. Greek brief pain inventory: validation and utility in cancer pain. Oncology. 2001;60(1):35-42. doi: 10.1159/000055294. PMID 11150906
- [Background] Mystakidou K, Tsilika E, Parpa E, Katsouda E, Galanos A, Vlahos L. The Hospital Anxiety and Depression Scale in Greek cancer patients: psychometric analyses and applicability. Support Care Cancer. 2004 Dec;12(12):821-5. doi: 10.1007/s00520-004-0698-y. Epub 2004 Oct 6. PMID 15480813
- [Background] Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2(3), 223-250. https://doi.org/10.1080/15298860309027
- [Background] O'Neill, L., Latchford, G., McCracken, L. M., & Graham, C. D. (2019). The development of the Acceptance and Commitment Therapy Fidelity Measure (ACT-FM): A delphi study and field test. Journal of Contextual Behavioral Science, 14, 111-118. https://doi.org/10.1016/j.jcbs.2019.08.008
- [Background] Roberts SB, Bonnici DM, Mackinnon AJ, Worcester MC. Psychometric evaluation of the Hospital Anxiety and Depression Scale (HADS) among female cardiac patients. Br J Health Psychol. 2001 Nov;6(Part 4):373-383. doi: 10.1348/135910701169278. PMID 12614511
- [Background] Smout, M., Davies, M., Burns, N., & Christie, A. (2014). Development of the valuing questionnaire (VQ). Journal of Contextual Behavioral Science, 3(3), 164-172. https://doi.org/10.1016/j.jcbs.2014.06.001
- [Background] Weis J, Tomaszewski KA, Hammerlid E, Ignacio Arraras J, Conroy T, Lanceley A, Schmidt H, Wirtz M, Singer S, Pinto M, Alm El-Din M, Compter I, Holzner B, Hofmeister D, Chie WC, Czeladzki M, Harle A, Jones L, Ritter S, Flechtner HH, Bottomley A; EORTC Quality of Life Group. International Psychometric Validation of an EORTC Quality of Life Module Measuring Cancer Related Fatigue (EORTC QLQ-FA12). J Natl Cancer Inst. 2017 May 1;109(5). doi: 10.1093/jnci/djw273. PMID 28376231
- [Background] Zacharia, M., Ioannou, M., Theofanous, A., Vasiliou, V. S., & Karekla, M. (2021). Does Cognitive Fusion show up similarly across two behavioral health samples? Psychometric properties and invariance of the Greek-Cognitive Fusion Questionnaire (G-CFQ). Journal of Contextual Behavioral Science. https://doi.org/10.1016/j.jcbs.2021.01.003
- [Background] Zettle, R. D., Gird, S. R., Webster, B. K., Carrasquillo-Richardson, N., Swails, J. A., & Burdsal, C. A. (2018). The Self-as-Context Scale: Development and preliminary psychometric properties. Journal of Contextual Behavioral Science, 10, 64-74. https://doi.org/10.1016/j.jcbs.2018.08.010
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- See also: ACThealthy Lab, University of Cyprus — https://www.ucy.ac.cy/acthealthy/en/